CLINICAL TRIAL: NCT03380637
Title: Ultrasound for Comparison of Gastric Volume in Pregnant Females Posted for Elective Lower Segment Cesarean Section With Non-pregnant Females Undergoing Elective Surgeries.
Brief Title: Ultrasound for Comparison of Gastric Antral Volume in Pregnants and Non-pregnants
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Snigdha Bellapukonda, Junior resident, MD Anesthesia, Department of Anesthesia and Intensive care, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 10565/PG-2Trg/2015/173-74
Record Dates: First submitted 2017-12-15; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Pregnancy
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant and non-pregnant females: The pregnant females posted for elective lower segment cesarean section and non-pregnant females posted for elective surgeries are scanned by ultrasound in the pre recovery room. The visibility of the gastric antrum is assessed. The qualitative and quantitative assessment is made and is compared.
  Interventions: Other: ultrasound

INTERVENTIONS:
Other: ultrasound — Sonosite ultrasound (Sonosite, FUJIFILM M-Turbo, made in USA)

SUMMARY:
This study evaluates the effectiveness of ultrasound in term pregnant patients posted for elective lower segment cesarean sections and compared them with non pregnant females posted for elective surgeries.

DETAILED DESCRIPTION:
There is increased risk of aspiration in pregnancy due to various reasons i.e. increased progesterone levels, decreased motilin levels and distortion of gastric antrum due to gravid uterus.Ultrasound was proposed to be point of care tool, to assess risk stomach. A comparison with respect to the effectiveness of ultrasound was made in this study. The visibility of gastric antrum by ultrasound in term pregnant females posted for elective lower segment cesarean sections was compared with non-pregnant females posted for elective surgeries.

The secondary aim of the study was to compare the gastric antrum in either groups qualitatively and quantitatively.

ELIGIBILITY:
Inclusion Criteria:Study group- Term pregnant patients, aged between 18 to 45 years, ASA II & III, having BMI between 18.5 to 30 kg/m2, scheduled for elective lower segment cesarean section.

Control group- Non-pregnant female patients, aged between 18 to 45 years, ASA I & II, having BMI between 18.5 to 30 kg/m2, scheduled for elective surgery.

Exclusion Criteria:Subjects with-

* Gastrointestinal pathology
* On any medication delaying gastric motility
* Systemic lupus erythematosis
* Diabetes mellitus
* Gestational diabetes
* Hypothyroidism Those who were not willing to give consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Term pregnant females posted for elective lower segment cesarean section and non-pregnant females posted for elective surgeries
Study Population: The study population are term pregnants posted for elective lower segment cesarean section and non-pregnant patients posted for elective surgeries in PGIMER.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2017-10-10 (Actual); Study Completion 2017-10-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness of ultrasound in pregnants and non-pregnants in terms of visibility | October 2016 to October 2017
  The effectiveness is stated in terms of percentage visibility and compared in pregnants and non-pregnants.

SECONDARY OUTCOMES:
Qualitative assessment of Gastric antrum | October 2016 to October 2017
  The qualitative grading is derived and is compared in the pregnants and non-pregnants.
Quantitative assessment of Gastric Antrum | October 2016 to October 2017
  The quantitative data is obtained from the derived formulae and is compared in pregnants and non-pregnants.

CONTACTS AND LOCATIONS:
Overall Officials: Snigdha Bellapukonda, MBBS, Principal Investigator — Post graduate institute of medical education and researchh

IPD SHARING:
Plan to Share IPD: Yes
Ultrasound for comparison of Gastric volume in pregnants undergoing Elective Lower Segment Cesarean Section and non-pregnant females undergoing elective surgeries.
Supporting Information: Study Protocol
Time Frame: December 2017 to December 2018
Access Criteria: public

REFERENCES:
- [Background] Perlas A, Davis L, Khan M, Mitsakakis N, Chan VW. Gastric sonography in the fasted surgical patient: a prospective descriptive study. Anesth Analg. 2011 Jul;113(1):93-7. doi: 10.1213/ANE.0b013e31821b98c0. Epub 2011 May 19. PMID 21596885